CLINICAL TRIAL: NCT00581776
Title: Phase II Study of VcR-CVAD With Rituximab Consolidation and Maintenance for Untreated Mantle Cell Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HO05401; 2011-0807 (Other: Institutional Review Board); A534260 (Other: UW Madison); SMPH\MEDICINE\HEM-ONC (Other: UW Madison)
Record Dates: First submitted 2007-12-19; First posted 2007-12-28 (Estimated); Results first posted 2011-02-15 (Estimated); Last update posted 2019-12-17 (Actual); Status verified 2016-05

CONDITIONS: Mantle Cell Lymphoma
Keywords: Untreated Mantle Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Mantle-Cell | interventions — Bortezomib; Rituximab; Cyclophosphamide; Doxorubicin; Vincristine; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- VCR-CVAD with rituximab maintenance (Experimental): Induction chemotherapy with Bortezomib, cyclophosphamide, rituximab, vincristine, doxorubicin, and dexamethasone. Subjects will receive 6 cycles of induction chemotherapy, of 21 days each. After completing induction, subjects will receive rituximab consolidation (4 weeks), and then rituximab maintenance therapy for up to 5 years.
  Interventions: Drug: Bortezomib; Drug: Rituximab; Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Vincristine; Drug: Dexamethasone

INTERVENTIONS:
Drug: Bortezomib — Administered by IV at 1.3 mg/m2 days 1 and 4 of each 21 day cycle.
  Other Names: Velcade, PS-341
Drug: Rituximab — Administered by IV 375 mg/m2 IV day 1 of each cycle during induction chemotherapy, then weekly for four weeks during consolidation therapy; and then once every 12 weeks for up to 5 years (or until disease progression).
  Other Names: Rituxan
Drug: Cyclophosphamide — Administered by IV at 300 mg/m2, 6 doses spaced 12 hours apart on days 1-3 of each cycle, to start after completion of rituximab infusion
  Other Names: cytoxan
Drug: Doxorubicin — Given as a continuous infusion, 50 mg/m2 over 48 hours days 1-2 of each cycle, to start after completion of rituximab infusion.
Drug: Vincristine — 1 mg administered by IV on day 3 of each cycle.
Drug: Dexamethasone — 40 mg orally on days 1-4 of each cycle.

SUMMARY:
Patients will receive Rituximab, Bortezomib, cyclophosphamide, Doxorubicin, Vincristine, Dexamethasone in three week intervals for 6 cycles; then rituximab consolidation (weekly x 4) , then one dose of rituximab every 12 weeks until 5 years or disease progression.

DETAILED DESCRIPTION:
Primary objective is to estimate the overall response rate (ORR) and the complete response rate (CRR) to the VcR CVAD regimen (response rate at completion of induction). Patients will receive Rituximab, Bortezomib, cyclophosphamide, Doxorubicin, Vincristine, Dexamethasone in three week intervals for 6 cycles; then rituximab consolidation (weekly x 4) , then one dose of rituximab every 12 weeks until 5 years or disease progression.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed CD20+ mantle cell lymphoma, with measurable or evaluable disease, no prior chemotherapy, immunotherapy or radiotherapy except for 1 cycle of CHOP-like chemotherapy.

Exclusion Criteria:

* Patients with known CNS disease, known HIV infection, grade 2 or greater peripheral neuropathy, history of myocardial infarction in last 6 months, or patients who are Hepatitis B Surface Antigen positive.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2005-05; Primary Completion 2012-11 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brad S Kahl, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University Of Wisconsin Cancer Center, Madison, Wisconsin, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | VCR-CVAD With Rituximab Maintenance
Started | 30
Completed | 27 (3 subjects did not complete the planned induction chemotherapy.)
Not Completed | 3
Not completed — Disease progression or no response | 3

BASELINE CHARACTERISTICS:
Arm/Group | VCR-CVAD With Rituximab Maintenance
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 22
  >=65 years | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 61 (26)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 24
Region of Enrollment [Number; unit: participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR) at the Completion of Induction Chemotherapy, Which is the Percent of Complete Responses (CR) Plus Percent of Partial Responses (PR).
Description: Patients were considered evaluable for response if they completed at least 2 cycles of therapy and had undergone an initial response evaluation, or had disease progression after 1 cycle of therapy.
  1999 International Working Group criteria defines a CR as patients with complete disappearance of disease, or regression of all lymph nodes to 1.5 cm in greatest diameter or less. Partial Response indicates patients responded to treatment with a reduction in the amount of tumor (50 percent or more). Overall response rate is the percent of complete responses plus the percent of partial responses.
Time Frame: At completion of induction therapy (21 weeks)
Measure: Number (95% Confidence Interval); unit: Percent of participants
Arm/Group | VCR-CVAD With Rituximab Maintenance
Number analyzed (Participants) | 30
Percent of participants | 90 [73 to 98]

2. Primary Outcome: Complete Response Rate (CR) at the End of Induction Chemotherapy
Description: Complete Response Rate (CRR) as defined by 1999 International Working Group criteria, is defined as patients with complete disappearance of disease, or regression of all lymph nodes to 1.5 cm in greatest diameter or less. All subjects who had completed 2 cycles of therapy and had at least one disease evaluation, or had completed 1 cycle of therapy with progressive disease, were considered evaluable.
Time Frame: at 21 weeks
Measure: Number (95% Confidence Interval); unit: percent of participants
Arm/Group | VCR-CVAD With Rituximab Maintenance
Number analyzed (Participants) | 30
percent of participants | 77 [73 to 98]

3. Secondary Outcome: 3 Year Progression Free Survival
Description: This is the percent of subjects who had not had any recurrence or relapse of disease as of 3 years after enrollment in the study.
Time Frame: 36 months
Measure: Number (95% Confidence Interval); unit: percent of participants
Arm/Group | VCR-CVAD With Rituximab Maintenance
Number analyzed (Participants) | 30
percent of participants | 63 [48 to 83]

4. Secondary Outcome: 3 Year Overall Survival (OS)
Description: This is the percent of participants who were still alive at 3 years after study entry.
Time Frame: 36 months
Measure: Number (95% Confidence Interval); unit: Percent of participants
Arm/Group | VCR-CVAD With Rituximab Maintenance
Number analyzed (Participants) | 30
Percent of participants | 86 [75 to 100]

ADVERSE EVENTS:
Time Frame: Adverse Event collection with 42 months median follow up
Arm/Group | VCR-CVAD With Rituximab Maintenance
Serious Adverse Events (participants affected / at risk) | 18/30
Other Adverse Events (participants affected / at risk) | 30/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | VCR-CVAD With Rituximab Maintenance (N=30)
Pain (Musculoskeletal and connective tissue disorders) | 1 (1) — Grade 3 pain, unrelated to investigational therapy
febrile neutropenia (Investigations) | 4 (4) — Febrile neutropenia
Infection (Infections and infestations) | 9 (9)
Dehydration Gr 3 (Gastrointestinal disorders) | 2 (2)
Creatinine Gr 2 (Renal and urinary disorders) | 1 (1)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Mucositis - Esophagitis (Gastrointestinal disorders) | 1 (1)
Thrombus (Cardiac disorders) | 2 (2) — 1 event of picc line clot, one Pulmonary embolus
myelosuppression (Blood and lymphatic system disorders) | 2 (2)
progressive disease (General disorders) | 1 (1) — admission and death due to progressive lymphoma
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | VCR-CVAD With Rituximab Maintenance (N=30)
Thrombocytopenia Gr 3 or 4 (Investigations) | 23
Neutropenia gr 3 or 4 (Investigations) | 20
Hemoglobin gr 3 (Investigations) | 8
Febrile Neutropenia gr 3 (Injury, poisoning and procedural complications) | 5
Infection with neutropenia (Infections and infestations) | 2
Infection without neutropenia (Infections and infestations) | 4
Hyperglycemia gr 3 (Investigations) | 4
hyponatremia gr 3 (Investigations) | 4
Hypophosphatemia gr 3 (Investigations) | 1
Dehydration gr 3 (Gastrointestinal disorders) | 2
Pulmonary Embolism Gr 4 (Cardiac disorders) | 1
Esophagitis Gr 3 (Gastrointestinal disorders) | 1
Mood alteration Gr 3 (Nervous system disorders) | 1
Pain gr 3 (Nervous system disorders) | 2
Sensory neuropathy gr 3 and 4 (Nervous system disorders) | 9
Fatigue gr 3 (General disorders) | 2
hypogammaglobulinemia (Immune system disorders) | 12/22
Infections secondary to hypogammaglobulinemia in maintenance therapy (Infections and infestations) | 6/22 (9)
delayed neutropenia during rituximab maintenance (Investigations) | 5/22 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less